CLINICAL TRIAL: NCT04763265
Title: A Double-Blinded, Randomized, Controlled Study to Compare the Efficacy, Time to Onset, and Duration of Effect of Botulinum Type A Toxins in the Treatment of Glabellar Frown Lines
Brief Title: Study to Compare 2 Botulinum Type A Toxins in the Treatment of Glabellar Frown Lines
Acronym: H2H
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Croma-Pharma GmbH (Industry)
Collaborators: Hugel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPH-201-201461
Record Dates: First submitted 2021-01-25; First posted 2021-02-21 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2021-01

CONDITIONS: Frown Lines

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized, double-blind, comparator-controlled study. The study will take place in the EU, US and Canada. The benefit of participation in this study is the expected reduction in the severity of glabellar frown lines. All subjects will benefit from free medical screenings and follow up.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Eligible subjects will be randomized at Baseline (Day 0) to Group A or B in a 1:1 randomization scheme. Investigators and subjects will be blinded to the treatment administered and will evaluate the severity of glabellar lines independently. The subjects should perform their assessment independently and ideally before the investigator, to ensure they are not biased by the investigator. The same investigator must complete the Baseline assessments and FWS at Week 4 (primary endpoint assessments) for a given subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (n=100): BoNT/A-DP (20 U, 0.5 mL) (Active Comparator): The injection sites should be prepared according to standard clinical procedures..
  A volume of 0.5 mL of the properly reconstituted BoNT/A-DP should be drawn into the sterile syringe and any air bubbles in the syringe barrel expelled. The needle used to reconstitute the product should be removed and replaced with a sterile insulin or tuberculin-type syringe of 1 mL volume with 0.01 mL graduation and with the gauge range of 30 to 33 G, which the investigator routinely uses for toxin administration.
  Each subject will receive a total of five i.m. injections of 4 U/0.1 mL (total of 20 U).
  Interventions: Biological: Botulinum toxin A "BoNT/A-DP"
- Group B (n=100): Botox Cosmetic (20 U, 0.5 mL) (Active Comparator): The injection sites should be prepared according to standard clinical procedures.
  A volume of 0.5 mL of the properly reconstituted Botox Cosmetic should be drawn into the sterile syringe and any air bubbles in the syringe barrel expelled. The needle used to reconstitute the product should be removed and replaced with a sterile insulin or tuberculin-type syringe of 1 mL volume with 0.01 mL graduation and with the gauge range of 30 to 33 G, which the investigator routinely uses for toxin administration.
  Each subject will receive a total of five i.m. injections of 4 U/0.1 mL (total of 20 U).
  Interventions: Biological: Botulinum toxin A "Botox Cosmetics"

INTERVENTIONS:
Biological: Botulinum toxin A "BoNT/A-DP" — To assess the efficacy of treatment with BoNT/A-DP in reducing the severity of glabellar frown lines at maximum frown.
  Arms: Group A (n=100): BoNT/A-DP (20 U, 0.5 mL)
Biological: Botulinum toxin A "Botox Cosmetics" — To assess the efficacy of treatment with Botox Cosmetics in reducing the severity of glabellar frown lines at maximum frown.
  Arms: Group B (n=100): Botox Cosmetic (20 U, 0.5 mL)

SUMMARY:
The purpose of the study is to provide preliminary comparative data on BoNT/A-DP versus Botox Cosmetic. Subsequently the sample size is primarily based on clinical judgement and practical considerations.

DETAILED DESCRIPTION:
This will be a multi-center, randomized, double-blind, comparator-controlled study. The study will take place in the EU, US and Canada.

To allow all subjects to profit from treatment and to obtain adequate data for BoNT/A DP treatment, the study will be comprised of a double-blinded treatment comparing BoNT/A-DP with Botox Cosmetic (ratio 1:1). Primary and secondary endpoints will compare efficacy, safety and subject satisfaction after a single treatment of the investigational BoNT/A DP to an existing commercially available product (Botox Cosmetic).

Two hundred subjects will be enrolled, which should allow for a precise estimate of response rate and for post-hoc sensitivity analyses.

The duration of study participation for each subject will be up to 18 weeks, to include screening (maximum of 2 weeks; re-screening will not be permitted), and a single treatment (comprised of one injection at five injection points) of BoNT/A-DP (Group A) or Botox Cosmetic (Group B) followed by six efficacy and safety follow-up visits. A total of 200 subjects will be randomized 1:1 to Group A or Group B at Baseline. Both investigators and subjects will be blinded to treatment. Investigators and subjects will evaluate the severity of glabellar lines independently.

ELIGIBILITY:
Inclusion Criteria:• Has moderate to severe glabellar frown lines at maximum frown (severity score of 2 or 3 on GLS-I/GLS-S) as determined by in clinic assessments by both the investigator and the subject (where: 0='none', 1='mild', 2='moderate', 3='severe').

* Subject has a stable medical condition with no uncontrolled systemic disease.
* Female subjects of childbearing potential must test negative for pregnancy and agree to use highly effective birth control during the course of the study.
* Subjects who wear glasses must be able to adequately self-assess the severity of their glabellar lines (according to the GLS-S), without glasses obstructing the forehead area.

Exclusion Criteria:

* Previous treatment with any serotype of botulinum toxin for any indication within the 12 months prior to Screening, or any planned treatment with botulinum toxin of any serotype for any reason during the study (other than the investigational treatment).
* Known hypersensitivity to either study medication or its excipients.
* Any medical condition that may place the subject at increased risk due to exposure to botulinum toxin, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, profound atrophy or weakness in the target muscles, or any other condition (at the investigator's discretion) that might interfere with neuromuscular function or contraindicate botulinum toxin therapy.
* Facial laser or light treatment, microdermabrasion, superficial peels or retinoid therapy within the three months prior to Screening or planned during the study.

  o Apart from the procedures specified above, previous treatment with any facial aesthetic procedure in the glabellar area (including chemical peeling, injection with biodegradable fillers, photo rejuvenation) within 12 months prior to Screening or planned during the study.
* Previous insertion of permanent material in the glabellar area, or planned insertion during the study.
* Any planned or history of surgery in the glabellar area and/or canthal line area, or scars in the glabellar and/or canthal line.
* Active skin disease/infection or irritation at the treatment area.
* Inability to substantially lessen glabellar frown lines and or lateral canthal lines even by physically spreading them apart.
* Use of a muscle relaxant within 2 weeks prior to Screening, or planned use during the study.
* Marked facial asymmetry or ptosis of eyelid and/or eyebrow, or current facial palsy or neuromuscular junction disorders as judged by the investigator.
* Pregnant, breastfeeding or planning to become pregnant during the study.
* Use of prohibited medication including anticholinergic drugs, or drugs which could interfere with neuromuscular function, including aminoglycoside antibiotics and curare-like compounds within 2 weeks prior to Screening or planned during the study.
* Planned surgery with general anesthetic (use of local anesthetic outside the glabellar area is permitted).
* Participation in another clinical study within one month of Screening and throughout the study.
* Previous participation in another botulinum toxin aesthetic study, which involved the treatment of glabellar, lines in combination with canthal lines and/or forehead lines in the previous 18 months.
* Chronic drug or alcohol abuse (as per investigator discretion).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - ATS Clinical Research, Santa Monica, California
  - Skin Research Institute LLC, Coral Gables, Florida
- Monika Sulovsky, Vienna, Austria
- Canada (2):
  - Institute Of Cosmetic, Oakville, Ontario
  - Sweat Clinics of Canada, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 208 enrolled participants, 200 met inclusion criteria and were randomized to treatment.
Groups:
- Group A (n=100): BoNT/A-DP (20 U, 0.5 mL): The injection sites should be prepared according to standard clinical procedures..
  A volume of 0.5 mL of the properly reconstituted BoNT/A-DP should be drawn into the sterile syringe and any air bubbles in the syringe barrel expelled. The needle used to reconstitute the product should be removed and replaced with a sterile insulin or tuberculin-type syringe of 1 mL volume with 0.01 mL graduation and with the gauge range of 30 to 33 G, which the investigator routinely uses for toxin administration.
  Each subject will receive a total of five i.m. injections of 4 U/0.1 mL (total of 20 U).
  Botulinum toxin A "BoNT/A-DP": To assess the efficacy of treatment with BoNT/A-DP in reducing the severity of glabellar frown lines at maximum frown.
- Group B (n=100): Botox Cosmetic (20 U, 0.5 mL): The injection sites should be prepared according to standard clinical procedures.
  A volume of 0.5 mL of the properly reconstituted Botox Cosmetic should be drawn into the sterile syringe and any air bubbles in the syringe barrel expelled. The needle used to reconstitute the product should be removed and replaced with a sterile insulin or tuberculin-type syringe of 1 mL volume with 0.01 mL graduation and with the gauge range of 30 to 33 G, which the investigator routinely uses for toxin administration.
  Each subject will receive a total of five i.m. injections of 4 U/0.1 mL (total of 20 U).
  Botulinum toxin A "Botox Cosmetics": To assess the efficacy of treatment with Botox Cosmetics in reducing the severity of glabellar frown lines at maximum frown.
Period: Overall Study
Arm/Group | Group A (n=100): BoNT/A-DP (20 U, 0.5 mL) | Group B (n=100): Botox Cosmetic (20 U, 0.5 mL)
Started | 100 | 100
Completed | 97 | 95
Not Completed | 3 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The population consists of all randomized subjects who had a baseline visit and at least one post-dose in-clinic assessment with the 4-point Facial Wrinkle Scale by either the investigator or the subject at Weeks 1, 2, or 4.
Groups:
- Group A: BoNT/A-DP (20 U, 0.5 mL): The injection sites should be prepared according to standard clinical procedures..
  A volume of 0.5 mL of the properly reconstituted BoNT/A-DP should be drawn into the sterile syringe and any air bubbles in the syringe barrel expelled. The needle used to reconstitute the product should be removed and replaced with a sterile insulin or tuberculin-type syringe of 1 mL volume with 0.01 mL graduation and with the gauge range of 30 to 33 G, which the investigator routinely uses for toxin administration.
  Each subject will receive a total of five i.m. injections of 4 U/0.1 mL (total of 20 U).
  Botulinum toxin A "BoNT/A-DP": To assess the efficacy of treatment with BoNT/A-DP in reducing the severity of glabellar frown lines at maximum frown.
- Group B: Botox Cosmetic (20 U, 0.5 mL): The injection sites should be prepared according to standard clinical procedures.
  A volume of 0.5 mL of the properly reconstituted Botox Cosmetic should be drawn into the sterile syringe and any air bubbles in the syringe barrel expelled. The needle used to reconstitute the product should be removed and replaced with a sterile insulin or tuberculin-type syringe of 1 mL volume with 0.01 mL graduation and with the gauge range of 30 to 33 G, which the investigator routinely uses for toxin administration.
  Each subject will receive a total of five i.m. injections of 4 U/0.1 mL (total of 20 U).
  Botulinum toxin A "Botox Cosmetics": To assess the efficacy of treatment with Botox Cosmetics in reducing the severity of glabellar frown lines at maximum frown.
- Total: Total of all reporting groups
Arm/Group | Group A: BoNT/A-DP (20 U, 0.5 mL) | Group B: Botox Cosmetic (20 U, 0.5 mL) | Total
Number analyzed (Participants) | 99 | 100 | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 90 | 92 | 182
  >=65 years | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (11.36) | 48.1 (12.04) | 48.5 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 86 | 172
  Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 21 | 39
  Not Hispanic or Latino | 81 | 79 | 160
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 87 | 90 | 177
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 39 | 34 | 73
  Austria | 22 | 23 | 45
  United States | 38 | 43 | 81
Fitzpatrick Skintype [Count of Participants; unit: Participants] — The Fitzpatrick skin type is a scale that classifies skin based on its reaction to sun exposure, specifically its tendency to burn or tan. It includes six types:
  Type I: very pale white skin, burns without tanning; Type II: white skin, burns and does not tan easily; Type III: fair skin, burns first then tans; Type IV: light brown skin, burns a little and tans easily; Type V: brown skin, easily tans to a darker color and rarely burns; Type VI: dark brown or black skin, never burns but tans darker
  Participants
    Type I | 2 | 5 | 7
    Type II | 33 | 32 | 65
    Type III | 31 | 32 | 63
    Type IV | 27 | 27 | 54
    Type V | 3 | 2 | 5
    Type VI | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Facial Wrinkle Scale (FWS) Score of 0 or 1 and an Improvement of ≥ 1 Points in FWS Score (at Maximum Frown) at Week 4 Visit Relative to Baseline, Based on Both the Investigators´ and the Subjects´ In-clinic Assessments.
Description: The primary endpoint is the percentage of subjects among BoNT/A-DP and Botox Cosmetic groups with a Facial Wrinkle Scale (FWS) score of 0 or 1 and an improvement of ≥ 1 points in FWS score (at maximum frown) at week 4 visit (of the first treatment cycle) relative to baseline (responders), based on both the investigators' and the subjects' in-clinic assessments. Thus, the primary endpoint is a composite endpoint comprising investigator and subject assessments of treatment effectiveness. FWS scores are a four-point rating scale as follows: 0 = no facial wrinkles; 1 = mild facial wrinkles; 2 = moderate facial wrinkles; and 3 = severe facial wrinkles. Subjects with missing in-clinic assessments with the FWS at Baseline or Week 4 were assigned as non-responders.
Time Frame: week 4
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: BoNT/A-DP (20 U, 0.5 mL) | Group B: Botox Cosmetic (20 U, 0.5 mL)
Number analyzed (Participants) | 99 | 100
Participants
  Responder based on Investigator's In-clinic Assessment | 95 | 97
  Responder based on Subject's In-clinic Assessment | 81 | 88

2. Secondary Outcome: Responder Status (With a Facial Wrinkle Scale (FWS) Score of 0 or 1 and at Least 1 Point Reduction at Maximum Frown) Based on Independent Investigator Assessment and Subject Assessment at Weeks 1, 2, 8, 12 and 16
Description: The percentage of responders based on the independent investigator assessment and subject assessment at Weeks 1, 2, 8, 12 and 16 after a single treatment with BoNT/A-DP and compared to a single treatment of Botox Cosmetic. Responder is defined as having a Facial Wrinkle Scale (FWS) score of 0 or 1 and at least 1 point reduction in FWS score at maximum frown over Baseline, on the 4-point FWS. FWS scores are ranked as 0 (no facial wrinkles), 1 (mild facial wrinkles), 2 (moderate facial wrinkles) and 3 (severe facial wrinkles). Subjects with missing in-clinic assessments with the FWS at Baseline or the respective visit were assigned as non-responders.
Time Frame: Weeks 1, 2, 8, 12 and 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: BoNT/A-DP (20 U, 0.5 mL) | Group B: Botox Cosmetic (20 U, 0.5 mL)
Number analyzed (Participants) | 99 | 100
Participants
  Responder Rate at Week 1 based on Investigator's In-clinic Assessment | 93 | 90
  Responder Rate at Week 1 based on Subject's In-clinic Assessment | 80 | 83
  Responder Rate at Week 2 based on Investigator's In-clinic Assessment | 93 | 95
  Responder Rate at Week 2 based on Subject's In-clinic Assessment | 83 | 91
  Responder Rate at Week 8 based on Investigator's In-clinic Assessment | 84 | 89
  Responder Rate at Week 8 based on Subject's In-clinic Assessment | 60 | 76
  Responder Rate at Week 12 based on Investigator's In-clinic Assessment | 66 | 78
  Responder Rate at Week 12 based on Subject's In-clinic Assessment | 43 | 56
  Responder Rate at Week 16 based on Investigator's In-clinic Assessment | 47 | 61
  Responder Rate at Week 16 based on Subject's In-clinic Assessment | 35 | 46

3. Secondary Outcome: Responder Status (With a Facial Wrinkle Scale (FWS) Score of 0 or 1 and at Least 2 Point Reduction at Maximum Frown) Based on Independent Investigator Assessment and Subject Assessment at Weeks 1, 2, 4, 8, 12 and 16
Description: The percentage of responders based on the independent investigator assessment and subject assessment at Weeks 1, 2, 4, 8, 12 and 16 after a single treatment with BoNT/A-DP and compared to a single treatment of Botox Cosmetic. Responder is defined as having a Facial Wrinkle Scale (FWS) score of 0 or 1 and at least 2 point reduction in FWS score at maximum frown over Baseline, on the 4-point FWS. FWS scores are ranked as 0 (no facial wrinkles), 1 (mild facial wrinkles), 2 (moderate facial wrinkles) and 3 (severe facial wrinkles). Subjects with missing in-clinic assessments with the FWS at Baseline or the respective visit were assigned as non-responders.
Time Frame: Weeks 1, 2, 4, 8, 12 and 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: BoNT/A-DP (20 U, 0.5 mL) | Group B: Botox Cosmetic (20 U, 0.5 mL)
Number analyzed (Participants) | 99 | 100
Participants
  Responder Rate at Week 1 based on Investigator's In-clinic Assessment | 80 | 79
  Responder Rate at Week 1 based on Subject's In-clinic Assessment | 68 | 72
  Responder Rate at Week 2 based on Investigator's In-clinic Assessment | 83 | 86
  Responder Rate at Week 2 based on Subject's In-clinic Assessment | 75 | 83
  Responder Rate at Week 4 based on Investigator's In-clinic Assessment | 82 | 88
  Responder Rate at Week 4 based on Subject's In-clinic Assessment | 67 | 81
  Responder Rate at Week 8 based on Investigator's In-clinic Assessment | 64 | 70
  Responder Rate at Week 8 based on Subject's In-clinic Assessment | 44 | 65
  Responder Rate at Week 12 based on Investigator's In-clinic Assessment | 37 | 52
  Responder Rate at Week 12 based on Subject's In-clinic Assessment | 27 | 39
  Responder Rate at Week 16 based on Investigator's In-clinic Assessment | 22 | 33
  Responder Rate at Week 16 based on Subject's In-clinic Assessment | 18 | 32

4. Secondary Outcome: Responder Status (With a Facial Wrinkle Scale (FWS) Score of 0 or 1 and at Least 1 Point Reduction at Rest) Based on Independent Investigator Assessment and Subject Assessment at Weeks 1, 2, 4, 8, 12 and 16
Description: The percentage of responders based on the independent investigator assessment and subject assessment at Weeks 1, 2, 4, 8, 12 and 16 after a single treatment with BoNT/A-DP and compared to a single treatment of Botox Cosmetic. Responder is defined as having a Facial Wrinkle Scale (FWS) score of 0 or 1 and at least 1 point reduction in FWS score at rest over Baseline, on the 4-point FWS. FWS scores are ranked as 0 (no facial wrinkles), 1 (mild facial wrinkles), 2 (moderate facial wrinkles) and 3 (severe facial wrinkles). Subjects with missing in-clinic assessments with the FWS at Baseline or the respective visit were assigned as non-responders.
Time Frame: Weeks 1, 2, 4, 8, 12 and 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: BoNT/A-DP (20 U, 0.5 mL) | Group B: Botox Cosmetic (20 U, 0.5 mL)
Number analyzed (Participants) | 99 | 100
Participants
  Responder Rate at Week 1 based on Investigator's In-clinic Assessment | 57 | 53
  Responder Rate at Week 1 based on Subject's In-clinic Assessment | 58 | 58
  Responder Rate at Week 2 based on Investigator's In-clinic Assessment | 65 | 64
  Responder Rate at Week 2 based on Subject's In-clinic Assessment | 70 | 64
  Responder Rate at Week 4 based on Investigator's In-clinic Assessment | 67 | 68
  Responder Rate at Week 4 based on Subject's In-clinic Assessment | 68 | 70
  Responder Rate at Week 8 based on Investigator's In-clinic Assessment | 63 | 62
  Responder Rate at Week 8 based on Subject's In-clinic Assessment | 57 | 60
  Responder Rate at Week 12 based on Investigator's In-clinic Assessment | 58 | 53
  Responder Rate at Week 12 based on Subject's In-clinic Assessment | 45 | 48
  Responder Rate at Week 16 based on Investigator's In-clinic Assessment | 45 | 52
  Responder Rate at Week 16 based on Subject's In-clinic Assessment | 36 | 48

5. Secondary Outcome: Time to Onset of Effect Based on Independent Investigator Assessment and Subject Assessment
Description: Time to onset of effect in days, as measured at Weeks 1, 2, and 4, based on independent investigator and subject assessments after a single treatment with BoNT/A-DP and compared to Botox Cosmetic. Onset of effect is defined as at least 1 point improvement in Glabellar Line Scale - Investigator (GLS-I) and Glabellar Line Scale - Subject (GLS-S) score relative to Baseline at maximum frown in glabellar lines. GLS-I and GLS-S both use the same 4-point scale, ranked as 0 (No lines/minimal lines), 1 (Mild lines), 2 (Moderate lines) and 3 (Severe lines).
Time Frame: From treatment at Day 0 to Week 4
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Group A: BoNT/A-DP (20 U, 0.5 mL) | Group B: Botox Cosmetic (20 U, 0.5 mL)
Number analyzed (Participants) | 99 | 100
Days | 8.0 [7.0 to 9.0] | 8.0 [7.5 to 8.0]

6. Secondary Outcome: Duration of Effect Based on Independent Investigator Assessment and Subject Assessment
Description: For subjects who are responders at week 4, duration of effect in days is assessed based on independent investigator and subject assessments after a single treatment with BoNT/A-DP and compared to Botox Cosmetic. Responder is defined as having a Facial Wrinkle Scale (FWS) score of 0 or 1 and at least 1 point reduction in FWS score at maximum frown over Baseline, on the 4-point FWS. FWS scores are ranked as 0 (no facial wrinkles), 1 (mild facial wrinkles), 2 (moderate facial wrinkles) and 3 (severe facial wrinkles). Effect is deemed to be lost when scores return to Baseline or worse values. Duration of effect is defined as (the date that loss of response occurred) - (date of single study treatment ) + 1.
Time Frame: 16 Weeks
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Group A: BoNT/A-DP (20 U, 0.5 mL) | Group B: Botox Cosmetic (20 U, 0.5 mL)
Number analyzed (Participants) | 99 | 100
Days
  Duration of effect for responders at Week 4 based on Investigator's in-clinic assessment: number analyzed (Participants) | 95 | 97
  Duration of effect for responders at Week 4 based on Investigator's in-clinic assessment | 132 [117 to 132] | NA [119 to NA] — Since more than 50% of subjects were still responders at Week 16, it was not possible to calculate the median or the upper limit of the 95% Confidence Interval for the median.
  Duration of effect for responders at Week 4 based on Subject's in-clinic assessment: number analyzed (Participants) | 81 | 88
  Duration of effect for responders at Week 4 based on Subject's in-clinic assessment | 116 [114 to 121] | NA [117 to NA] — Since more than 50% of subjects were still responders at Week 16, it was not possible to calculate the median or the upper limit of the 95% Confidence Interval for the median.

7. Secondary Outcome: FACE-Q Satisfaction With Outcome Scale Based on Subject Assessment at Weeks 4, 12 and 16 Satisfaction With Outcome Scale.
Description: Summary of FACE-Q satisfaction with outcome scale based on subject assessment at weeks 4, 12 and 16 after a single treatment and compared to Botox Cosmetic. The FACE-Q Satisfaction with Outcome scale is a patient-reported outcome measure designed to assess a patient's satisfaction with the results of a facial aesthetic procedure. This scale comprises six items, each with four response options: "definitely agree," "somewhat agree," "somewhat disagree," and "definitely disagree."
Time Frame: Weeks 4, 12 and 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: BoNT/A-DP (20 U, 0.5 mL) | Group B: Botox Cosmetic (20 U, 0.5 mL)
Number analyzed (Participants) | 99 | 100
Participants
  Week 4 - pleased: Definitely disagree | 2 | 0
  Week 4 - pleased: Somewhat disagree | 3 | 3
  Week 4 - pleased: Somewhat agree | 17 | 12
  Week 4 - pleased: Definitely agree | 77 | 84
  Week 4 - pleased: Missing | 0 | 1
  Week 4 - expected: Definitely disagree | 4 | 0
  Week 4 - expected: Somewhat disagree | 5 | 6
  Week 4 - expected: Somewhat agree | 33 | 34
  Week 4 - expected: Definitely agree | 57 | 59
  Week 4 - expected: Missing | 0 | 1
  Week 4 - great: Definitely disagree | 2 | 1
  Week 4 - great: Somewhat disagree | 8 | 7
  Week 4 - great: Somewhat agree | 23 | 15
  Week 4 - great: Definitely agree | 66 | 76
  Week 4 - great: Missing | 0 | 1
  Week 4 - look in the mirror: Definitely disagree | 1 | 1
  Week 4 - look in the mirror: Somewhat disagree | 12 | 8
  Week 4 - look in the mirror: Somewhat agree | 31 | 30
  Week 4 - look in the mirror: Definitely agree | 55 | 60
  Week 4 - look in the mirror: Missing | 0 | 1
  Week 4 - fantastic: Definitely disagree | 4 | 3
  Week 4 - fantastic: Somewhat disagree | 13 | 11
  Week 4 - fantastic: Somewhat agree | 25 | 18
  Week 4 - fantastic: Definitely agree | 57 | 67
  Week 4 - fantastic: Missing | 0 | 1
  Week 4 - miraculous: Definitely disagree | 11 | 4
  Week 4 - miraculous: Somewhat disagree | 16 | 19
  Week 4 - miraculous: Somewhat agree | 32 | 27
  Week 4 - miraculous: Definitely agree | 40 | 49
  Week 4 - miraculous: Missing | 0 | 1
  Week 12 - pleased: Definitely disagree | 10 | 3
  Week 12 - pleased: Somewhat disagree | 6 | 7
  Week 12 - pleased: Somewhat agree | 28 | 24
  Week 12 - pleased: Definitely agree | 50 | 60
  Week 12 - pleased: Missing | 5 | 6
  Week 12 - expected: Definitely disagree | 11 | 6
  Week 12 - expected: Somewhat disagree | 11 | 9
  Week 12 - expected: Somewhat agree | 29 | 33
  Week 12 - expected: Definitely agree | 43 | 46
  Week 12 - expected: Missing | 5 | 6
  Week 12 - great: Definitely disagree | 9 | 5
  Week 12 - great: Somewhat disagree | 14 | 12
  Week 12 - great: Somewhat agree | 28 | 22
  Week 12 - great: Definitely agree | 43 | 55
  Week 12 - great: Missing | 5 | 6
  Week 12 - look in the mirror: Definitely disagree | 13 | 4
  Week 12 - look in the mirror: Somewhat disagree | 14 | 15
  Week 12 - look in the mirror: Somewhat agree | 33 | 36
  Week 12 - look in the mirror: Definitely agree | 34 | 39
  Week 12 - look in the mirror: Missing | 5 | 6
  Week 12 - fantastic: Definitely disagree | 12 | 7
  Week 12 - fantastic: Somewhat disagree | 22 | 18
  Week 12 - fantastic: Somewhat agree | 27 | 27
  Week 12 - fantastic: Definitely agree | 33 | 42
  Week 12 - fantastic: Missing | 5 | 6
  Week 12 - miraculous: Definitely disagree | 25 | 8
  Week 12 - miraculous: Somewhat disagree | 14 | 27
  Week 12 - miraculous: Somewhat agree | 31 | 30
  Week 12 - miraculous: Definitely agree | 24 | 29
  Week 12 - miraculous: Missing | 5 | 6
  Week 16 - pleased: Definitely disagree | 12 | 5
  Week 16 - pleased: Somewhat disagree | 10 | 8
  Week 16 - pleased: Somewhat agree | 21 | 20
  Week 16 - pleased: Definitely agree | 54 | 62
  Week 16 - pleased: Missing | 2 | 5
  Week 16 - expected: Definitely disagree | 12 | 6
  Week 16 - expected: Somewhat disagree | 14 | 12
  Week 16 - expected: Somewhat agree | 31 | 31
  Week 16 - expected: Definitely agree | 40 | 46
  Week 16 - expected: Missing | 2 | 5
  Week 16 - great: Definitely disagree | 10 | 8
  Week 16 - great: Somewhat disagree | 20 | 13
  Week 16 - great: Somewhat agree | 20 | 18
  Week 16 - great: Definitely agree | 47 | 56
  Week 16 - great: Missing | 2 | 5
  Week 16 - look in the mirror: Definitely disagree | 12 | 11
  Week 16 - look in the mirror: Somewhat disagree | 20 | 15
  Week 16 - look in the mirror: Somewhat agree | 29 | 30
  Week 16 - look in the mirror: Definitely agree | 36 | 39
  Week 16 - look in the mirror: Missing | 2 | 5
  Week 16 - fantastic: Definitely disagree | 17 | 10
  Week 16 - fantastic: Somewhat disagree | 19 | 17
  Week 16 - fantastic: Somewhat agree | 24 | 21
  Week 16 - fantastic: Definitely agree | 37 | 47
  Week 16 - fantastic: Missing | 2 | 5
  Week 16 - miraculous: Definitely disagree | 26 | 14
  Week 16 - miraculous: Somewhat disagree | 14 | 20
  Week 16 - miraculous: Somewhat agree | 35 | 33
  Week 16 - miraculous: Definitely agree | 22 | 28
  Week 16 - miraculous: Missing | 2 | 5

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious AEs (SAEs) and AEs of Special Interest (AESIs)
Description: Frequency, seriousness and severity of treatment-emergent adverse events (TEAEs), serious AEs (SAEs) and AEs of special interest (AESIs), as well as causal relationship to the study medication and the study procedure, during the entire study period. A subject with multiple occurrences of an adverse event is counted only once within the worst severity category.
Time Frame: through study completion, an average of 16 weeks
Population: The population consists of all subjects who received at least one injection with the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: BoNT/A-DP (20 U, 0.5 mL) | Group B: Botox Cosmetic (20 U, 0.5 mL)
Number analyzed (Participants) | 100 | 100
Participants
  Subjects with any treatment-emergent adverse events | 25 | 22
  Subjects with any serious treatment-emergent adverse events | 0 | 1
  Subjects with any treatment-emergent adverse events of special interest | 0 | 1
  Subjects with any severe treatment-emergent adverse events | 0 | 0
  Subjects with any moderate treatment-emergent adverse events | 5 | 4
  Subjects with any mild treatment-emergent adverse events | 20 | 18
  Subjects with any treatment-emergent adverse events related to study medication | 4 | 3
  Subjects with any treatment-emergent adverse events related to study procedure | 6 | 8

9. Secondary Outcome: Change From Baseline in Blood Pressure at Weeks 1, 4, 12 and 16
Description: Summary of change from baseline in diastolic/systolic blood pressure at weeks 1, 4, 12 and 16 after a single treatment and compared to Botox Cosmetic.
Time Frame: Weeks 1, 4, 12, and 16
Population: The population consists of all subjects who received at least one injection with the study medication. Only subjects with available data at the respective visit were analyzed.
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A: BoNT/A-DP (20 U, 0.5 mL) | Group B: Botox Cosmetic (20 U, 0.5 mL)
Number analyzed (Participants) | 100 | 100
millimeters of mercury
  Diastolic Blood Pressure (mmHg) - Week 1 - Change from Baseline: number analyzed (Participants) | 99 | 98
  Diastolic Blood Pressure (mmHg) - Week 1 - Change from Baseline | 0.9 (8.48) | -1.9 (8.50)
  Diastolic Blood Pressure (mmHg) - Week 4 - Change from Baseline: number analyzed (Participants) | 99 | 99
  Diastolic Blood Pressure (mmHg) - Week 4 - Change from Baseline | 0.1 (8.29) | -1.9 (8.80)
  Diastolic Blood Pressure (mmHg) - Week 12 - Change from Baseline: number analyzed (Participants) | 90 | 92
  Diastolic Blood Pressure (mmHg) - Week 12 - Change from Baseline | -0.1 (9.64) | -1.2 (10.19)
  Diastolic Blood Pressure (mmHg) - Week 16 - Change from Baseline: number analyzed (Participants) | 95 | 86
  Diastolic Blood Pressure (mmHg) - Week 16 - Change from Baseline | 1.0 (9.30) | -1.6 (10.85)
  Systolic Blood Pressure (mmHg) - Week 1 - Change from Baseline: number analyzed (Participants) | 99 | 98
  Systolic Blood Pressure (mmHg) - Week 1 - Change from Baseline | 0.2 (10.84) | -2.4 (12.29)
  Systolic Blood Pressure (mmHg) - Week 4 - Change from Baseline: number analyzed (Participants) | 99 | 99
  Systolic Blood Pressure (mmHg) - Week 4 - Change from Baseline | 0.3 (11.44) | -0.9 (12.78)
  Systolic Blood Pressure (mmHg) - Week 12 - Change from Baseline: number analyzed (Participants) | 90 | 92
  Systolic Blood Pressure (mmHg) - Week 12 - Change from Baseline | 0.6 (11.79) | -1.3 (14.77)
  Systolic Blood Pressure (mmHg) - Week 16 - Change from Baseline: number analyzed (Participants) | 95 | 86
  Systolic Blood Pressure (mmHg) - Week 16 - Change from Baseline | 1.5 (12.30) | -1.5 (15.52)

10. Secondary Outcome: Change From Baseline in Pulse Rate at Weeks 1, 4, 12 and 16
Description: Summary of change from baseline in pulse rate at weeks 1, 4, 12 and 16 after a single treatment and compared to Botox Cosmetic.
Time Frame: Weeks 1, 4, 12, and 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Group A: BoNT/A-DP (20 U, 0.5 mL) | Group B: Botox Cosmetic (20 U, 0.5 mL)
Number analyzed (Participants) | 100 | 100
beats/min
  Pulse Rate (beats/min) - Week 1 - Change from Baseline: number analyzed (Participants) | 99 | 98
  Pulse Rate (beats/min) - Week 1 - Change from Baseline | 2.2 (10.25) | -0.4 (9.94)
  Pulse Rate (beats/min) - Week 4 - Change from Baseline: number analyzed (Participants) | 99 | 99
  Pulse Rate (beats/min) - Week 4 - Change from Baseline | 1.0 (11.60) | 1.6 (9.46)
  Pulse Rate (beats/min) - Week 12 - Change from Baseline: number analyzed (Participants) | 90 | 92
  Pulse Rate (beats/min) - Week 12 - Change from Baseline | 1.2 (11.72) | -0.2 (11.90)
  Pulse Rate (beats/min) - Week 16 - Change from Baseline: number analyzed (Participants) | 95 | 86
  Pulse Rate (beats/min) - Week 16 - Change from Baseline | 1.9 (11.02) | 0.5 (11.31)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Group A (n=100): BoNT/A-DP (20 U, 0.5 mL) | Group B (n=100): Botox Cosmetic (20 U, 0.5 mL)
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 1/100
Other Adverse Events (participants affected / at risk) | 11/100 | 15/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (n=100): BoNT/A-DP (20 U, 0.5 mL) (N=100) | Group B (n=100): Botox Cosmetic (20 U, 0.5 mL) (N=100)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (n=100): BoNT/A-DP (20 U, 0.5 mL) (N=100) | Group B (n=100): Botox Cosmetic (20 U, 0.5 mL) (N=100)
Corona virus infection (Infections and infestations) | 2 (2) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Viral test positive (Investigations) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 6 (6) | 10 (11)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/65/NCT04763265/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT04763265/SAP_001.pdf